CLINICAL TRIAL: NCT03566277
Title: Project Step: Evaluating Deposit Contracts and Daily Feedback to Promote Walking in Overweight and Obese Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Drexel University (Other)
Collaborators: Psi Chi (Other); Qualtrics (Unknown); American College of Sports Medicine (Other)
Responsible Party: Principal Investigator, Stephanie Kerrigan, Doctoral Candidate, Drexel University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1601004185-1
Record Dates: First submitted 2018-06-12; First posted 2018-06-25 (Actual); Last update posted 2018-06-25 (Actual); Status verified 2018-06

CONDITIONS: Physical Activity; Sedentary Lifestyle; Obesity; Overweight
MeSH Terms: conditions — Motor Activity; Sedentary Behavior; Obesity; Overweight | interventions — Blood Glucose Self-Monitoring; Fertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single-arm trial (Experimental): All participants will undergo each of three conditions during the study.
  Interventions: Behavioral: Self-monitoring; Behavioral: Incentives; Behavioral: Feedback

INTERVENTIONS:
Behavioral: Self-monitoring — Participants will have access to a wrist-worn activity monitor and have a daily step goal
Behavioral: Incentives — Participants will have a deposit contract, wherein they will lose money if a goal is not reached, or double their money if a goal is reached
Behavioral: Feedback — Participants will receive text message feedback each day about progress towards their goal

SUMMARY:
The purpose of this study is to test whether deposit contracts, wherein individuals invest their own money with the study to serve as the incentive, with or without daily feedback about progress help individuals to increase step counts and more often meet a step goal compared to self-monitoring only.

DETAILED DESCRIPTION:
Approximately 68% of adults are overweight or obese, which is associated with increased risk for health conditions, including cardiovascular disease, type 2 diabetes, and cancer. These individuals are more often sedentary than the general population, which compounds the risk for these same conditions. While the benefits of engaging in physical activity are well-established, few individuals are able to successfully increase activity to recommended levels. Existing intervention programs, often derived from theories such as social cognitive theory or related theories, have had limited success. Behavioral economics offers a promising alternative, suggesting that engagement in any behavior is based on the maximizing utility and happiness. Interventions based on this theory aim to increase the immediate benefit of engaging in physical activity, often using a financial incentive.

This study will last for 16 weeks. Each participant will invest $42 with the study, and be exposed to to each of three interventions. All participants will have the use of a FitBit for ongoing self-monitoring and a step-count goal of 10,000 steps per day. In one condition, these will be the only interventions you receive. In one condition, you will receive a monetary consequence for meeting or not meeting the goal. Each day during the incentive conditions, you will be eligible to lose $0.75 of your own money for not meeting the goal, or to earn back $0.75 of your money plus $0.75 from the study (i.e., a total of $1.50) for meeting the goal. In the third condition, you will have daily feedback mid-afternoon about your distance from the goal and the money you stand to gain or lose. You will be made aware of what condition you are in.

ELIGIBILITY:
Inclusion Criteria:

* 25 kg/m2 ≤ BMI ≤ 45 kg/m2
* Age 18-70
* Currently inactive (engages in less than 6,000 steps/day on at least 4 of 7 days per week, confirmed by FitBit at baseline)
* Able to engage in moderate amount of walking
* Able to receive email/text messages from study staff

Exclusion Criteria:

- medical or psychiatric conditions that would make it difficult to comply with study protocols

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2016-12-01 (Actual); Primary Completion 2017-08-01 (Actual); Study Completion 2017-08-08 (Actual)

PRIMARY OUTCOMES:
Step counts | Throughout 16-week study, measured as the average of each two-week block (i.e., each time condition changes)
  Daily number of steps taken
Goal attainment | Throughout 16-week study, measured as the average of each two-week block (i.e., each time condition changes)
  Proportion of days step goal was met

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kerrigan SG, Forman EM, Patel M, Williams D, Zhang F, Crosby RD, Butryn ML. Evaluating the Feasibility, Acceptability, and Effects of Deposit Contracts With and Without Daily Feedback to Promote Physical Activity. J Phys Act Health. 2020 Jan 1;17(1):29-36. doi: 10.1123/jpah.2018-0589. PMID 31698334